CLINICAL TRIAL: NCT01977872
Title: JointADventure: A Worksite Activity-Diet Intervention for Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Rowland W. Chang, Professor of Preventive Medicine, Medicine, and Physical Medicine & Rehabilitation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AR062317 (NIH); R21AR062317 (NIH)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Knee Pain; Osteoarthritis, Knee
Keywords: Arthritis; Physical Activity; Diet
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A worksite activity-diet intervention (Experimental): A 12 month intensive program that includes individual sessions, interactive group sessions and online activities.
  Interventions: Behavioral: A worksite activity-diet intervention
- Motiva Program (No Intervention): The Motiva Program is the internal corporate wellness program offered to all BCBSIL employees.

INTERVENTIONS:
Behavioral: A worksite activity-diet intervention
  Arms: A worksite activity-diet intervention

SUMMARY:
JointADventure: A worksite activity-diet intervention for chronic knee pain is a randomized controlled trial evaluation of a physical activity and nutritional worksite intervention to decrease symptoms and disability associated with knee osteoarthritis (OA), a major public health problem and a leading cause of work disability and work absenteeism/presenteeism in the US workforce.

The overarching goal of this project is to find an effective and sustainable intervention strategy that can assist large populations of persons with or at risk for knee OA to attain and maintain healthy dietary and physical activity behaviors. This project has to potential to have a tremendous impact on improving symptoms and quality of life of persons with chronic knee pain and decreasing the functional limitation, work absenteeism/presenteeism, and soaring healthcare utilization associated with knee OA.

DETAILED DESCRIPTION:
We will utilize a partnership with Blue Cross Blue Shield of Illinois (BCBSIL), a highly supportive wellness partner, with a strong history of investment in the health of its employees and subscribers. The combined Activity/Dietary (AD) intervention is administered by health professionals trained in motivational interviewing as healthy lifestyle coaches.

Over the first 6 months, the coaches provide:

* individualized counseling based on a comprehensive assessment of baseline clinical, functional and behavioral factors that are barriers to healthy physical activity and dietary behaviors
* group education, the content of which is modeled after the highly successful Diabetes Prevention Program physical activity/dietary intervention, and customized for those with knee symptoms.

Follow-up assessments continue for 6 additional months.

Specific aims are to:

1. assess the feasibility of conducting a randomized controlled trial of the JointADventure intervention at this worksite
2. estimate the effectiveness of the intervention to decrease body weight, improve dietary habits, and increase objectively-measured physical activity
3. to improve objectively measured functional performance
4. to improve self-reported arthritis-specific and generic health status and health utility

ELIGIBILITY:
Inclusion Criteria:

* BCBSIL employee
* Must be able to ambulate household distances (50 ft)
* Must be able to read and speak English
* Pain, aching, stiffness in or around one or both knees on most days for at least one month during the past 12 months
* BMI of >25, but <40

Exclusion Criteria:

* Primary diagnosis of fibromyalgia
* Any co-morbidity that is more functionally limiting than the knee symptoms (e.g. spinal stenosis, peripheral vascular disease or residual effects of stroke)
* Comorbid condition (based on medication review) that contraindicates a physical activity or dietary intervention
* Total joint replacement surgery within 1 year or plans for total joint replacement in the next 12 months
* Plans to relocate away from the Chicago-land area in the next 12 months
* Being on a special diet that is inconsistent with the DASH diet
* Concurrent involvement in a weight loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change in accelerometer counts/day | Baseline, 3, 6 and 12 months
change in kilocalorie intake | Baseline, 3, 6 and 12 months
percent change in body weight | Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
20 meter walk | Baseline, 3, 6 and 12 months
  Change in walking velocity
chair stand test | Baseline, 3, 6 and 12 months
  Change in chair-stand rate

OTHER OUTCOMES:
Quality of Life | Baseline, 3 months, 6 months, 12 months
  Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)pain and function scores, Patient-Reported Objective Measurement Information System (PROMIS)scores, and change in Short Form 6D (SF-6D) utility scores

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Blue Cross Blue Shield of Illinois, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine Department of Preventive Medicine, Chicago, Illinois